CLINICAL TRIAL: NCT04447534
Title: Does Zinc Supplementation Enhance the Clinical Efficacy of Chloroquine/Hydroxychloroquine in Treatment of COVID-19?
Brief Title: Zinc With Chloroquine/Hydroxychloroquine in Treatment of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tanta zinc chloroquine
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: COVID
MeSH Terms: interventions — Chloroquine; Hydroxychloroquine; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroquine or hydroxychloroquine (Experimental): Chloroquine or hydroxychloroquine alone
  Interventions: Drug: Chloroquine or hydroxychloroquine
- Chloroquine or hydroxychloroquine with zinc (Experimental): Chloroquine or hydroxychloroquine with zinc
  Interventions: Drug: Chloroquine or hydroxychloroquine; Drug: zinc

INTERVENTIONS:
Drug: Chloroquine or hydroxychloroquine — Chloroquine or hydroxychloroquine
  Other Names: alexoquine, chloroquine, hydroquine
Drug: zinc — Zinc tablets
  Arms: Chloroquine or hydroxychloroquine with zinc

SUMMARY:
we want to investigate if zinc supplementation enhance the clinical efficacy of chloroquine in treatment of COVID-19.

DETAILED DESCRIPTION:
we want to investigate if zinc supplementation enhance the clinical efficacy of chloroquine in treatment of COVID-19. As, zinc may be of value in these cases and may be of value in enhancing chloroquine effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive COVID-19.

Exclusion Criteria:

* Contraindications or hypersensitivity to chloroquine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with improvement or mortality | 2 weeks
  The number of patients with improvement or mortality.

CONTACTS AND LOCATIONS:
Overall Officials: sherief Abd-Elsalam, Ass. Prof., Principal Investigator — ass. Prof. Tropical Medicine
Locations (1):
- Tanta university hospital, Assuit University, Ainshams University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd-Elsalam S, Soliman S, Esmail ES, Khalaf M, Mostafa EF, Medhat MA, Ahmed OA, El Ghafar MSA, Alboraie M, Hassany SM. Do Zinc Supplements Enhance the Clinical Efficacy of Hydroxychloroquine?: a Randomized, Multicenter Trial. Biol Trace Elem Res. 2021 Oct;199(10):3642-3646. doi: 10.1007/s12011-020-02512-1. Epub 2020 Nov 27. PMID 33247380